CLINICAL TRIAL: NCT07296861
Title: HomeGrown: A Family-based Lifestyle Intervention to Support Healthy Development of Young Children With Down Syndrome
Acronym: HomeGrown
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 25-2418; R01DK128174 (NIH)
Record Dates: First submitted 2025-12-18; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Down Syndrome; Child Obesity
Keywords: home environmental
MeSH Terms: conditions — Down Syndrome; Pediatric Obesity | interventions — Waiting Lists

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1- HomeGrown program (Experimental): Participants will receive interventions.
  Interventions: Behavioral: The HomeGrown
- Arm 2 Waitlist control (Active Comparator): Participants will receive interventions after study completion, 6-month delayed start.
  Interventions: Other: Waitlist

INTERVENTIONS:
Behavioral: The HomeGrown — The implementation model for supporting home environment changes focuses on engaging families in Homegrown, giving them access to interactive online tools and resources that guide behavior change, and providing monthly support check-in calls as they work to adopt evidence-based healthy eating and physical activity practices at home. Families will participate in the 6-month program with support from a trained health educator. The HomeGrown program begins with a family orientation session, followed by access to the HomeGrown web application.
  Participants will have access to HomeGrown intervention which is a 6-month program that helps families improve healthy eating and physical activity at home. Families start with an orientation session, then use the HomeGrown web application with interactive tools and resources. Monthly check-in calls with a trained health educator provide guidance and support throughout the program.
  Arms: Arm 1- HomeGrown program
Other: Waitlist — Participants will have a 1-hour training with the interventionist to learn how to use a website (not HomeGrown). Access to HomeGrown will be provided after the 6-month study is completed.
  Arms: Arm 2 Waitlist control

SUMMARY:
The goal of this project is to evaluate an adapted health promotion program, HomeGrown, designed to improve the health of young children with Down syndrome by supporting families in making healthy home environmental changes. There is a significant need for evidence-based programs that address healthy eating and physical activity within this population, as most existing interventions have been developed for typically developing children. By tailoring the program to the unique needs of families of young children with Down syndrome, this project aims to advance inclusion and equity in health behavior promotion.

This R61/R33 study will assess the feasibility (R61 Phase) and subsequent efficacy (R33 Phase) of the HomeGrown program in improving family practices related to nutrition and physical activity. During the R61 feasibility phase, 38 primary caregivers of children aged 2-6 years with Down syndrome will be enrolled in a 6-month randomized controlled trial. Families will be randomized 1:1 to either the HomeGrown intervention or a waitlist control group (6-month delayed start), stratified by the child's biological sex (male/female) and age (2-3 vs. 4-6 years). All measures will be collected at baseline and at 6-month follow-up.

The R61 feasibility phase will address three specific aims:

Accrual: Achieve an enrollment rate of 10 families per month, supporting feasibility for the R33 efficacy phase.

Engagement: Demonstrate that families use at least 70% of available HomeGrown intervention components, measured using the digital behavior change interventions engagement scale.

Data Collection & Retention: Achieve at least 80% retention with completion of all outcome assessments.

By addressing key gaps in nutrition and physical activity research for young children with Down syndrome, this study has the potential to improve health outcomes for an underserved population and inform future clinical and community health promotion efforts.

ELIGIBILITY:
Inclusion Criteria:

Adult:

* Ability to provide informed consent
* 18 years or older
* Primary caregiver of a child with Down syndrome aged 2 to 6 years old
* Have access to WI-FI or smartphone
* Be able to read and speak English

Children:

* Be 2-6 years old.
* Are diagnosed with Down syndrome
* Are not reliant on tube feeding

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Accrual Rate | Baseline
  Percent of eligible participants who agreed to join study.
Participant Engagement | 6 months
  Digital behavior change engagement scale will be measured as number of participants completed digital intervention.
Participant Retention | 6 months
  Percent of participants who completed 6-month measures.

SECONDARY OUTCOMES:
Child Physical Activity | 6 months
  GT3X+ accelerometers (ActiGraph, Pensacola, FL) are small wearable devices that measure movement and physical activity levels. worn on children's waist for 7 consecutive days. Reminders about wearing and returning the device will be sent via email/text throughout each assessment period. Video instructions will also be available through the web application. Accelerometer data will be used to calculate the number of minutes participants spend in each physical activity level (sedentary, light, moderate, vigorous, and total non-sedentary).
Child Diet Quality | 6 months
  Caregivers will complete 24-hour dietary recalls to report their child's food and beverage intake using the Automated Self-Administered 24-hour (ASA24) Dietary Assessment Tool. Caregivers will receive a standardized email with login details, instructions, and a prompt to complete the recall, followed by a reminder text on their assigned recall days. If a recall is still not completed, data collectors will make a final attempt to complete it with the caregiver by phone.
  Using the ASA24 output, Healthy Eating Index-Toddlers-2020 (HEI-2020) scores will be calculated. The HEI-2020 reflects how closely a child's diet aligns with dietary guidelines, with scores ranging from 0 to 100; higher scores indicate better diet quality.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Willis, PhD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- UNC Center for Health Promotion and Disease Prevention, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual, de-identified data will be shared in compliance with NIH data sharing policies. They will be shared via the funding institute's required INCLUDE Data Coordinating Center as well as UNC Dataserve.

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials